CLINICAL TRIAL: NCT03861078
Title: The Effect of Electronic Cigarette Liquid Characteristics in Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM20015258; U54DA036105 (NIH); F31DA047018 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-03-04 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cigarette smokers (Experimental): Each participant will participate in 5 sessions. During each session, participants will complete a 10-puff, directed product use bout, and then have the option later to puff as little or as much as they like during a 30-minute self administration task.
  Session 1: Own brand cigarette use Session 2: ECIG 15 mg nicotine, sweetened Session 3: ECIG Lab Session ECIG 15 mg nicotine, unsweetened Session 4: ECIG Lab Session ECIG 0 mg nicotine, sweetened Session 5: ECIG Lab Session ECIG 0 mg nicotine, unsweetened
  Interventions: Other: Own Brand Cigarette; Other: ECIG 15 mg nicotine, sweetened; Other: ECIG 15 mg nicotine, unsweet; Other: ECIG 0 mg nicotine, sweetened; Other: ECIG 0 mg nicotine, unsweet

INTERVENTIONS:
Other: Own Brand Cigarette — Effects of own brand cigarette use.
Other: ECIG 15 mg nicotine, sweetened — Effects of using a 30 Watt ECIG filled with 15 mg nicotine, sweetened liquid
Other: ECIG 15 mg nicotine, unsweet — Effects of using a 30 Watt ECIG filled with 15 mg nicotine, unsweet liquid
Other: ECIG 0 mg nicotine, sweetened — Effects of using a 30 Watt ECIG filled with 0 mg nicotine, sweetened liquid
Other: ECIG 0 mg nicotine, unsweet — Effects of using a 30 Watt ECIG filled with 0 mg nicotine, unsweet liquid

SUMMARY:
The purpose of this study is to determine differences in nicotine delivery, user behaviors, subjective effects, and physiological effects, when cigarette smokers use an electronic cigarette with different nicotine (and sweetener) concentrations relative to using their own brand of cigarettes.

ELIGIBILITY:
Inclusion Criteria-- Participants must be:

* Healthy (determined by self-report)
* Between the ages of 21-55 years old
* Current cigarette smokers
* Wiling to provide informed consent
* Able to attend the lab session and abstain from tobacco/nicotine products as required
* Agree to use designated products according to the study protocol

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Individuals who weigh less than 110 pounds.

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Study Director — Virginia Commonwealth University
Locations (1):
- Clinical Behavioral Pharmacology Laboratory, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maloney SF, Hoetger C, Bono RS, Lester Scholtes R, Combs M, Karaoghlanian N, Lipato T, Breland A, Eissenberg T. Assessment of human abuse potential of an unflavored, sucralose-sweetened electronic cigarette in combustible cigarette smokers. Exp Clin Psychopharmacol. 2024 Oct;32(5):588-603. doi: 10.1037/pha0000720. Epub 2024 May 30. PMID 38815111

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant will participate in 5 sessions. Sessions differ by the tobacco product used (see study arms). The sessions are ordered by latin-square; however, session order was NOT expected to change any outcomes and order effects are not relevant to the study. Therefore all outcome data was merged and analyzed only by arm and session without regard to order.
Groups:
- Cigarette Smokers: Each participant will participate in 5 sessions. During each session, participants will complete a 10-puff, directed product use bout, and then have the option later to puff as little or as much as they like during a 30-minute self administration task.
  Session 1: Own brand cigarette use Session 2: ECIG 15 mg nicotine, sweetened Session 3: ECIG Lab Session ECIG 15 mg nicotine, unsweetened Session 4: ECIG Lab Session ECIG 0 mg nicotine, sweetened Session 5: ECIG Lab Session ECIG 0 mg nicotine, unsweetened
  Own Brand Cigarette: Effects of own brand cigarette use.
  ECIG 15 mg nicotine, sweetened: Effects of using a 30 Watt ECIG filled with 15 mg nicotine, sweetened liquid
  ECIG 15 mg nicotine, unsweet: Effects of using a 30 Watt ECIG filled with 15 mg nicotine, unsweet liquid
  ECIG 0 mg nicotine, sweetened: Effects of using a 30 Watt ECIG filled with 0 mg nicotine, sweetened liquid
  ECIG 0 mg nicotine, unsweet: Effects of using a 30 Watt ECIG filled with 0 mg nicotine, unsweet liquid
Period: Overall Study
Arm/Group | Cigarette Smokers
Started | 22
Session 1: Own Brand Cigarette Use | 14
Session 2: ECIG 15 mg Nicotine, Sweetened | 14
Session 3: ECIG Lab Session ECIG 15 mg Nicotine, Unsweetened | 14
Session 4: ECIG Lab Session ECIG 0 mg Nicotine, Sweetened | 14
Session 5: ECIG Lab Session ECIG 0 mg Nicotine, Unsweetened | 14
Completed | 14
Not Completed | 8
Not completed — COVID-19 shut down | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — lack of venous access | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.07 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 14.21 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration
Description: Change in plasma nicotine concentration. Changes in plasm nicotine concentration during puff bout are considered to be the more relevant and accurate values so analysis and results reporting will focus on change from baseline to immediately following 10-puff bout.
Time Frame: Blood will be taken 4 times in each session to examine changes from baseline (approx 70 minutes) to immediately following a ten-puff bout (approx 80 minutes), and immediately before (approx 140 minutes) and after the PRT (approx 180 minutes).
Population: One participant had incomplete blood data and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 13
ng/ml
  Own Brand | 12.32 (8.3)
  Unsweetened, 0 mg/ml nicotine | -0.22 (1.0)
  Unsweetened, 15 mg/ml nicotine | 7.09 (8.6)
  Sweetened, 15 mg/ml nicotine | 5.85 (7.0)
  Sweetened, 0 mg/ml nicotine | -0.29 (1.1)

2. Primary Outcome: Progressive Ratio Task - Breakpoint
Description: The progressive ratio task (PRT) is a self-administration task that will take 30-minutes to complete. It will begin by requiring ten computer key presses to earn the first puff of the session product, and this requirement will increase by 30% (i.e., 10, 13, 17, etc.) after each reinforcer (puff) is earned and consumed. The PRT will have three outcome measures (1) breakpoint (maximum number of key presses completed to earn a puff), (2) number of puffs, and (3) latency (sec) to initiate key pressing. Breakpoint is reported here.
Time Frame: This task will begin approximately an hour and ten minutes after the 10-puff directed product use bout.
Population: Cigarette smokers
Measure: Mean (Standard Deviation); unit: Key presses
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
Key presses
  Unsweetened, 0 mg/ml nicotine | 416.07 (502.0)
  Sweetened, 0 mg/ml nicotine | 307.29 (415.3)
  Unsweetened, 15 mg/ml nicotine | 336.43 (687.3)
  Sweetened, 15 mg/ml nicotine | 492.86 (811.0)
  Own brand cigarette | 812.86 (1132.3)

3. Secondary Outcome: Puff Volume
Description: The volume of each puff, in ml, averaged over the 10-puff use bout
Time Frame: Puff volume will be measured during the approximately 5-minute, 10-puff use bout.
Population: Cigarette smokers
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
ml
  Unsweetened, 0 mg/ml nicotine | 207.17 (124.5)
  Sweetened, 0 mg/ml nicotine | 233.47 (157.7)
  Unsweetened, 15 mg/ml nicotine | 130.57 (110.4)
  Sweetened, 15 mg/ml nicotine | 166.51 (141.0)
  Own brand cigarette | 65.12 (48.3)

4. Secondary Outcome: Puff Duration
Description: The duration of each puff, in seconds, averaged over the 10-puff use bout
Time Frame: The duration of each puff will be measured during the approximately 5-minute, 10-puff use bout.
Population: Cigarette smokers
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
seconds
  Unsweetened, 0 mg/ml nicotine | 2.54 (1.8)
  Sweetened, 0 mg/ml nicotine | 2.74 (1.5)
  Unsweetened, 15 mg/ml nicotine | 1.60 (0.7)
  Sweetened, 15 mg/ml nicotine | 1.94 (1.4)
  Own brand cigarette | 2.06 (1.3)

5. Other Pre Specified Outcome: Hughes-Hatsukami Questionnaire
Description: This scale will be used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0-100, with lower scores indicating less severe symptoms. There are no sub-scales. Items are analyzed separately.
Time Frame: This questionnaire will be administered 4 times in each session to examine changes from baseline (70 minutes) to immediately following a ten-puff bout (80 minutes), and immediately before (140 minutes) and after the PRT (180 minutes)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Positive and Negative Affect Schedule
Description: This scale will be used to measure positive and negative affect and consists of 20-items that are scored on a 5-point likert scale ranging from "very slightly or not at all" to "extremely". The items from this scale are scored into two dimensions: Positive Affect and Negative Affect.
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Drug Effects Questionnaire
Description: This questionnaire assess a respondent's feelings after recently using tobacco or nicotine products. It has a total of five items that participants rate from not at all to extremely scored 0-100. Each item is scored and analyzed separately (there are no sub-scales).
Time Frame: as for outcome 5
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Heart Rate
Description: Change in heart rate, measure in beats per minute.
Time Frame: Heart rate will be measured continuously throughout the session, and will be used to examine changes in HR from baseline (70 minutes) to during (75 minutes) and immediately following a ten-puff bout (80 minutes)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Inter Puff Interval
Description: The time between each puff, in seconds.
Time Frame: Inter puff interval will be measured during the approximately 5-minute, 10-puff use bout.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Flow Rate
Description: The rate of air flow during each puff, in ml/second.
Time Frame: Flow rate will be measured during the approximately 5-minute, 10-puff use bout.
Reporting Status: Not Posted

11. Primary Outcome: Progressive Ratio Task - Number of Puffs
Description: The progressive ratio task (PRT) is a self-administration task that will take 30-minutes to complete. It will begin by requiring ten computer key presses to earn the first puff of the session product, and this requirement will increase by 30% (i.e., 10, 13, 17, etc.) after each reinforcer (puff) is earned and consumed. The PRT will have three outcome measures (1) breakpoint (maximum number of key presses completed to earn a puff), (2) number of puffs, and (3) latency (sec) to initiate key pressing. Number of puffs is reported here.
Time Frame: This task will begin approximately an hour and ten minutes after the 10-puff directed product use bout.
Population: Cigarette smokers
Measure: Mean (Standard Deviation); unit: Number of puffs
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
Number of puffs
  Unsweetened, 0 mg/ml nicotine | 7.64 (4.2)
  Sweetened, 0 mg/ml nicotine | 6.21 (4.7)
  Unsweetened, 15 mg/ml nicotine | 5.07 (5.1)
  Sweetened, 15 mg/ml nicotine | 7.21 (5.0)
  Own brand cigarette | 9.93 (4.1)

12. Primary Outcome: Progressive Ratio Task - Latency
Description: The progressive ratio task (PRT) is a self-administration task that will take 30-minutes to complete. It will begin by requiring ten computer key presses to earn the first puff of the session product, and this requirement will increase by 30% (i.e., 10, 13, 17, etc.) after each reinforcer (puff) is earned and consumed. The PRT will have three outcome measures (1) breakpoint (maximum number of key presses completed to earn a puff), (2) number of puffs, and (3) latency (milliseconds) to initiate key pressing. Latency is reported here.
Time Frame: This task will begin approximately an hour and ten minutes after the 10-puff directed product use bout.
Population: Cigarette smokers
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cigarette Smokers
Number analyzed (Participants) | 14
milliseconds
  Unsweetened, 0 mg/ml nicotine | 161176.93 (473649.1)
  Sweetened, 0 mg/ml nicotine | 390300.43 (764004.4)
  Unsweetened, 15 mg/ml nicotine | 315803.79 (636134.5)
  Sweetened, 15 mg/ml nicotine | 263130.86 (651141.0)
  Own brand cigarette | 6500.64 (6972.8)

ADVERSE EVENTS:
Description: This protocol was minimal risk and All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Cigarette Smokers | ECIG 15 mg Nicotine, Sweetened | ECIG 15 mg Nicotine, Unsweet | ECIG 0 mg Nicotine, Sweetened | ECIG 0 mg Nicotine, Unsweet
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03861078/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03861078/ICF_000.pdf